

840 Walnut Street Philadelphia, PA 19107 215-928-3000 1-877-AT-WILLS www.willseye.org

An Educational Intervention to Increase Adoption of Selective Laser Trabeculoplasty as First-Line Treatment for Glaucoma

NCT03365778

Informed Consent Form for Ophthalmologists

July 11, 2017

PI: L. Jav Katz. MD

## Wills Eye Hospital An Educational Intervention to Increase Adoption of Selective Laser Trabeculoplasty as First-Line Treatment for Glaucoma

## **Study Consent Form**

| <u></u> |
|---|
| Participant Name: |
| We are asking you to participate in a research study. |
| This study is an educational intervention to understand opinions, knowledge and beliefs about the choice of glaucoma treatment, (specifically medication versus selective laser trabeculoplasty (SLT)) in patients diagnosed with glaucoma and to get input from the physician who offers such treatments. |
| If you voluntarily agree to participate, you will view an educational video before and after you are asked questions about your beliefs and attitudes about SLT as first line therapy in patients newly diagnosed with glaucoma. You will also be asked to complete an online survey regarding these views. |
| Although there may be no benefit to you to participate in the study, the results of this research study may be of help to other glaucoma patients and future ophthalmologists. This study will take approximately 30 minutes of your time. |
| There are no risks associated with participating in this study. |
| If you have questions about the study, contact research personnel at 215-928-3197. If you have questions about your rights as a research participant, contact the Wills Eye IRB at 215-928-3141. |
| Subject Signature: |
| Name of Person Obtaining Consent: |
| Signature of Person Obtaining Consent: |